CLINICAL TRIAL: NCT04596293
Title: A Randomised, Double-blind, Placebo-controlled Study of Orally Administered BBT-401-1S in Subjects With Moderate to Severe Ulcerative Colitis, Incorporating a Response-adaptive, Double-blind Extension Phase
Brief Title: Efficacy and Safety of Orally Administered BBT-401-1S in Subjects With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bridge Biotherapeutics, Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BBT401-UC-005
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BBT-401-1S (800mg) (Experimental): * Induction Phase: BBT-401 800mg for 8 weeks
  * Extension Phase: After 8 weeks,
    * Participants who achieved clinical remission in the induction phase will continue the same treatment for 8 weeks
    * Participants who did not achieve clinical remission in the induction phase will receive BBT-401 1600mg for 8 weeks
  Interventions: Drug: BBT-401-1S or Placebo
- BBT-401-1S (1,600mg) (Experimental): * Induction Phase: BBT-401 1600mg for 8 weeks
  * Extension Phase: After 8 weeks, Participants will continue the same treatment for 8 weeks
  Interventions: Drug: BBT-401-1S or Placebo
- Placebo (Placebo Comparator): * Induction Phase: Placebo for 8 weeks
  * Extension Phase: After 8 weeks,
    * Participants who achieved clinical remission in the induction phase will continue the same treatment for 8 weeks
    * Participants who did not achieve clinical remission in the induction phase will receive BBT-401 800mg for 8 weeks
  Interventions: Drug: BBT-401-1S or Placebo

INTERVENTIONS:
Drug: BBT-401-1S or Placebo — Administered by 200mg capsules of BBT-401-1S or placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled, proof of clinical principle study to explore the efficacy and safety of orally administered BBT-401-1S in subjects with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race, ≥18 and ≤60 years of age.
* Have been diagnosed with active UC for ≥3 months prior to Day 1, as determined by clinical and endoscopic evidence and documented in a histopathology evaluation.
* Have a total Mayo score ≥6, an endoscopic subscore ≥2, rectal bleeding subscore ≥1, and a stool frequency subscore ≥1, regardless of standard of care history.
* Able to comprehend and willing to voluntarily sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

* Have received:

  1. intravenous corticosteroids, rectally administered corticosteroids, or rectally administered 5-aminosalicylic acid within 3 weeks, or
  2. Janus kinase (JAK) inhibitors within 2 weeks, or
  3. cyclosporine, mycophenolate, tacrolimus, or methotrexate within 5 weeks, or
  4. anti-TNF-α biologics within 9 weeks, or
  5. any other biologics (including ustekinumab and vedolizumab) for the treatment of UC within 12 weeks.
* Have received orally administered azathioprine or 6-mercaptopurine that has been stable for <8 weeks.
* Have received orally administered 5-aminosalicylic acid, sulphasalazine, or low-dose corticosteroids (prednisolone ≤20 mg/day or equivalent) that have been stable for <5 weeks.
* Have received any other concomitant medications for UC that have been stable (ie, have not started dosing with a new drug or had a change to their dosing regimen) for <7 days or 5 half-lives, whichever is longer.
* Have Crohn's disease, indeterminate colitis, ischaemic colitis, fulminant colitis, toxic megacolon, chronic (as determined by the investigator) pancolitis, confined proctitis (distal, ≤15 cm), or symptomatic intestinal stenosis.
* Have a history of extensive colonic resection (subtotal or total colectomy) or are anticipated to require surgical intervention for UC.
* Have an ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
* Have a positive test for Clostridium difficile, or have evidence of treatment for Clostridium difficile infection or other pathogenic bowel infection within 60 days or for another intestinal pathogen within 30 days prior to Day 1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (9):
  - Premier Gastroenterology, Little Rock, Arkansas
  - Saini Surinder S MD, Fountain Valley, California
  - Gastro Care Institute, Lancaster, California
  - Intercity Gastroentertology, Fresh Meadows, New York
  - Javara Research, Charlotte, North Carolina
  - Inves Clinic, McAllen, Texas
  - Discovery Clinical Trials - AACT, Pflugerville, Texas
  - Velocity Clinical Research, Riverton, Utah
  - West Jordan, West Jordan, Utah
- Poland (4):
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - VITA LONGA Sp. z o.o., Katowice, Silesian Voivodeship
  - Centrum Medyczne Melita Medical, Wroclaw, Wroclaw
  - Uniwersytecki Szpital Kliniczny Nr. 1 im. Norberta Barlickiego, Lodz, Łódź Voivodeship
- South Korea (7):
  - Inje University Haeundae Paik Hospital, Haeundae, Busan Gwang'yeogsi
  - Kyungpook National University Chilgok Hospital, Bugok, Daegu
  - Wonju Severance Christian Hospital, Wŏnju, Gang'weondo
  - Yeungnam University Hospital, Daegu, Gwang'yeogsi
  - Korea University Ansan Hospital, Ansan, Gyeonggido
  - Inje University, Seoul Paik Hospital, Junggu, Seoul
  - The Catholic university of Korea, Seoul St Mary's Hospital, Seocho, Seoul Teugbyeolsi
- Ukraine (9):
  - Municipal Non-Profit Enterprise City Clinical Hospital No. 2 named after prof. O.O. Shalimov of the, Kharkiv, Kharkivs’ka Oblast’
  - Municipal Non-Profit Enterprise Kherson City Clinical Hospital named after E.E.Karabelesha of Kherso, Kherson, Kherson Oblast
  - Medical Centre of the Limited Liability Company Medical Clinic Blagomed, Treatment and Diagnostic Di, Kyiv, Kyïv
  - Communal Non-profit enterprise Kyiv City Clinical Hospital No. 18, of the executive body of the Kyiv, Kyiv, Kyïv
  - Medical Center RCLIN Ukraine of the Limited Liability Company Cardiocom, Obukhiv, Kyïv
  - Municipal Enterprise Volyn Regional Clinical Hospital of the Volyn Regional Council, Department of S, Luts'k, Vinnytsia Oblast
  - Communal Non-profit enterprise Vinnytsya city clinical hospital 1 gastroenterology department, Vinnytsia, Vinnytsia Oblast
  - Medical Center of LLC Oxford Medical-Vinnytsia, Vinnytsia, Vinnytsia Oblast
  - Municipal Non-Profit Enterprise of the Kyiv Regional Council Kyiv Regional Hospital, Therapeutics De, Kyiv

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with moderate to severe Ulcerative Colitis (UC) were to be randomly assigned in a 1:1:1 ratio to 1 of 3 treatment groups. A total of 38 participants were enrolled and evaluated as Safety Population. Out of 38 participants, and 33 were considered Intent-to-Treatment Population and evaluated for study outcomes.
Period: Induction Phase Week 0-8
Arm/Group | Placebo | BBT-401-1S (800mg) | BBT-401-1S (1,600mg)
Started | 11 | 11 | 11
Safety Population | 13 | 12 | 13
Completed | 11 | 11 | 10
Not Completed | 0 | 0 | 1
Period: Extension Phase Week 8-16
Arm/Group | Placebo | BBT-401-1S (800mg) | BBT-401-1S (1,600mg)
Started (One subject completed induction phase of BBT-401-1S 1600mg did not participated in extension phase.) | 11 | 11 | 9
Safety Population | 6 | 8 | 17
Completed | 11 | 10 | 8
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo for 8 weeks as induction phase + Placebo or BBT-401-1S 800mg for 8 weeks as extension phase
- BBT-401-1S (800mg): BBT-401-1S 800mg for 8 weeks as induction phase + BBT-401-1S 800mg or BBT-401-1S 1600mg for 8 weeks as extension phase
- BBT-401-1S (1,600mg): BBT-401-1S 1600mg for 8 weeks as induction phase + BBT-401-1S 1600mg for 8 weeks as extension phase
- Total: Total of all reporting groups
Arm/Group | Placebo | BBT-401-1S (800mg) | BBT-401-1S (1,600mg) | Total
Number analyzed (Participants) | 11 | 11 | 11 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (9.6) | 35.0 (9.9) | 42.1 (9.1) | 41.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 7 | 7 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 11 | 10 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 10 | 10 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 0 | 1 | 1 | 2
  United States | 0 | 0 | 1 | 1
  Ukraine | 11 | 6 | 8 | 25
  Poland | 0 | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Clinical Response by Total Mayo Score at Day 57
Description: Clinical Response was defined as a Total Mayo Score, as measured by a reduction of ≥ 3 points and ≥ 30% improvement from baseline of Total Mayo Score, which included a decrease in rectal bleeding subscore of ≥ 1 point or an absolute rectal bleeding subscore ≤ 1
Time Frame: Day 57
Population: The intent-to-treat (ITT) population included all subjects who receive at least 1 dose of study drug, and who have a partial Mayo score recorded on Day 1 and at least 1 post-baseline Mayo score recorded. Subjects are categorized in the treatment group to which they are randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | BBT-401-1S (800mg) | BBT-401-1S (1,600mg)
Number analyzed (Participants) | 11 | 11 | 11
Percentage of participants | 63.6 [30.8 to 89.1] | 54.5 [23.4 to 83.3] | 54.5 [23.4 to 83.3]
Statistical Analysis 1: Comparison: Placebo vs BBT-401-1S (800mg); Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: BBT-401-1S (800mg) vs BBT-401-1S (1,600mg); Test type: Other; p = 1.0000, Fisher Exact

2. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Remission by Total Mayo Score at Day 57
Description: Clinical Remission was defined as a Total Mayo score, as measured by a total Mayo score of ≤ 2 points, with no individual subscore exceeding 1 point. Change from baseline to Day 57 in Total Mayo Score. The Total Mayo Score is consisted of 4 subscores (stool frequency, rectal bleeding, findings on endoscopy, physician's global assessment), each graded from 0 to 3 with higher scores indicating more severe disease
Time Frame: Day 57
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | BBT-401-1S (800mg) | BBT-401-1S (1,600mg)
Number analyzed (Participants) | 11 | 11 | 11
Percentage of Participants | 36.4 [10.9 to 69.2] | 18.2 [2.3 to 51.8] | 9.1 [0.2 to 41.3]
Statistical Analysis 1: Comparison: Placebo vs BBT-401-1S (800mg); Test type: Other; p = 0.6351, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs BBT-401-1S (1,600mg); Test type: Other; p = 0.3108, Fisher Exact

3. Secondary Outcome: Percentage of Participants Who Achieved an Endoscopic Remission at Day 57
Description: Endoscopic Remission was defined as a Mayo endoscopic subscore of 0 or 1. Change from baseline to Day 57 in Total Mayo Score. The Total Mayo Score is consisted of 4 subscores (stool frequency, rectal bleeding, findings on endoscopy, physician's global assessment), each graded from 0 to 3 with higher scores indicating more severe disease
Time Frame: Day 57
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | BBT-401-1S (800mg) | BBT-401-1S (1,600mg)
Number analyzed (Participants) | 11 | 11 | 11
Percentage of Participants | 45.5 [16.7 to 76.6] | 36.4 [10.9 to 69.2] | 27.3 [6.0 to 61.0]
Statistical Analysis 1: Comparison: Placebo vs BBT-401-1S (800mg); Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs BBT-401-1S (1,600mg); Test type: Other; p = 0.6594, Fisher Exact

4. Secondary Outcome: Change From Baseline to Day 57 in Total Mayo Score
Description: Change from Baseline to Day 57 in Total Mayo Score. Change from baseline to Day 57 in Total Mayo Score. The Total Mayo Score, ranged from 0 to 12, are sum of 4 subscores. Subscores are stool frequency, rectal bleeding, findings on endoscopy, and physician's global assessment, each graded from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Baseline, Day 57
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | BBT-401-1S (800mg) | BBT-401-1S (1,600mg)
Number analyzed (Participants) | 11 | 11 | 11
Scores on a scale
  Baseline | 8.8 (1.08) | 9.1 (1.70) | 8.4 (1.75)
  Day 57 | 4.5 (3.17) | 6.2 (3.37) | 5.6 (2.55)
  Change from Baseline | -4.3 (2.72) | -2.9 (2.47) | -2.6 (1.71)
Statistical Analysis 1: Comparison: Placebo vs BBT-401-1S (800mg); Test type: Other; p = 0.5808, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs BBT-401-1S (1,600mg); Test type: Other; p = 0.2143, ANCOVA

ADVERSE EVENTS:
Time Frame: From ICF consent up to 16 weeks for those who had completed the study or discontinued early
Description: The safety population included all subjects who receive at least 1 dose of study drug. Subjects are categorized in the treatment group of the treatment they actually receive.
Groups:
- Placebo/Induction Phase: Participants who received placebo in induction phase for 8 weeks
- BBT-401-1S 800mg/Induction Phase: Participants who received BBT-401-1S 800mg in induction phase for 8 weeks
- BBT-401-1S 1600mg/Induction Phase: Participants who received BBT-401-1S 1600mg in induction phase for 8 weeks
- Placebo/Extension Phase: Participants who received placebo in extension phase for 8 weeks
- BBT-401-1S 800mg/ Extension Phase: Participants who received BBT-401-1S 800mg in extension phase for 8 weeks
- BBT-401-1S 1600mg/ Extension Phase: Participants who received BBT-401-1S 1600mg in extension phase for 8 weeks
Arm/Group | Placebo/Induction Phase | BBT-401-1S 800mg/Induction Phase | BBT-401-1S 1600mg/Induction Phase | Placebo/Extension Phase | BBT-401-1S 800mg/ Extension Phase | BBT-401-1S 1600mg/ Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/13 | 0/6 | 0/8 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/12 | 0/13 | 0/6 | 0/8 | 0/17
Other Adverse Events (participants affected / at risk) | 1/13 | 3/12 | 1/13 | 1/6 | 2/8 | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Induction Phase (N=13) | BBT-401-1S 800mg/Induction Phase (N=12) | BBT-401-1S 1600mg/Induction Phase (N=13) | Placebo/Extension Phase (N=6) | BBT-401-1S 800mg/ Extension Phase (N=8) | BBT-401-1S 1600mg/ Extension Phase (N=17)
Bartholin's cyst removal (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 — Term from vocabulary, MedDRA 23.1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Induction Phase (N=13) | BBT-401-1S 800mg/Induction Phase (N=12) | BBT-401-1S 1600mg/Induction Phase (N=13) | Placebo/Extension Phase (N=6) | BBT-401-1S 800mg/ Extension Phase (N=8) | BBT-401-1S 1600mg/ Extension Phase (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Term from vocabulary, MedDRA 23.1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 — Term from vocabulary, MedDRA 23.1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Term from vocabulary, MedDRA 23.1
Abscess drainage (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 — Term from vocabulary, MedDRA 23.1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Term from vocabulary, MedDRA 23.1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Term from vocabulary, MedDRA 23.1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Term from vocabulary, MedDRA 23.1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 — Term from vocabulary, MedDRA 23.1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Term from vocabulary, MedDRA 23.1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 — Term from vocabulary, MedDRA 23.1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 — Term from vocabulary, MedDRA 23.1
Coagulation factor decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 — Term from vocabulary, MedDRA 23.1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Term from vocabulary, MedDRA 23.1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 — Term from vocabulary, MedDRA 23.1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 — Term from vocabulary, MedDRA 23.1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Term from vocabulary, MedDRA 23.1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Term from vocabulary, MedDRA 23.1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Term from vocabulary, MedDRA 23.1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Term from vocabulary, MedDRA 23.1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Term from vocabulary, MedDRA 23.1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04596293/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT04596293/SAP_001.pdf